CLINICAL TRIAL: NCT05504512
Title: Feasible Surgical Treatment of Peripelvic Cyst by Percutaneous Nephroscopy
Brief Title: Percutaneous Nephroscopic Treatment of Parapelvic Cysts
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 202208180
Record Dates: First submitted 2022-08-14; First posted 2022-08-17 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-08

CONDITIONS: Kidney Stone; Parapelvic Cyst; Kidney Diseases; Recurrence
Keywords: Parapelvic Cyst; Recurrence; Kidney Diseases
MeSH Terms: conditions — Kidney Calculi; Kidney Diseases; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parapelvic cyst
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Background of the project: The surgical treatment of parapelvic cysts is currently less researched and there is no gold standard for surgery. Previously, in percutaneous nephrolithotomy, we found that fenestration and fenestration drainage in the simultaneous treatment of pararenal pelvis cysts under nephroscopic nephroscopic surgery has clear curative effect, less trauma, and quicker recovery.

Objective: To clarify the safety, efficacy and long-term efficacy of percutaneous nephroscopy in the treatment of parapelvic cysts.

Nature: Retrospective case cohort study. Basic research process: Retrospective collection of cases in our hospital who underwent percutaneous nephroscopy for the treatment of parapelvic cysts, and comparison of preoperative and postoperative cyst size changes and long-term efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Has undergone percutaneous nephroscopic surgery for parapelvic cysts
* Ability to receive study follow-up

Exclusion Criteria:

* Patient refuses or is unable to give consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone percutaneous nephroscopic surgery for parapelvic cysts
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-11-30 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
cyst size | At least 1 year after percutaneous nephroscopy for parapelvic cysts
  Cyst maximum plane diameter

CONTACTS AND LOCATIONS:
Overall Officials: Yu Cui, M.D., Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya hospital of central south university, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided